CLINICAL TRIAL: NCT05835973
Title: Evaluation of Sleep Changes as Early Markers of Relapse in Patients With Inflammatory Bowel Diseases (IBD).
Brief Title: Evaluation of Sleep Changes in Inflammatory Bowel Diseases (IBD) Patients.
Acronym: RECIDREAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0907
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Disease Bowel; Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Diseases; Crohn's disease; ulcerative colitis; sleep deprivation; relapse
MeSH Terms: conditions — Intestinal Diseases; Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases; Sleep Deprivation; Recurrence | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep activity (Experimental): Actigraphy : Patient will wear actinometers on the wrist for 1 year continuously. In the study, MotionWatch 8 actimeters will be used, a class 1 medical device with CE mark (EN ISO 13485:2016 standard). They will be provided by the company camntech.
  Ancillary Study:
  DREEM 3 headband : a subgroup of patients will wear the headband during 2 nights every 3 months.
  Interventions: Other: Sleep activity; Other: Questionnaires

INTERVENTIONS:
Other: Sleep activity — Actinography : Patient will wear actinometers on the wrist for 1 year continuously. In the study, MotionWatch 8 actimeters will be used, a class 1 medical device with CE mark (EN ISO 13485:2016 standard).
  Ancillary study :
  DREEM 3 headband : a subgroup of patients will wear the headband during 2 nights every 3 months.
Other: Questionnaires — The PSQI, EPWORTH, FACIT-F, ISI, and ICSD-3 questionnaires will be completed by patients every 3 months during their follow-up consultation according to the usual management.
  The questionnaire by Horne and Ostberg will be completed by the patients only during the inclusion visit.

SUMMARY:
Inflammatory Bowel Diseases (IBD) go through two phases: flare and remission. Prediction of flares and identification of patients in remission but at high risk of flare are a major issue when taking care of IBD patients.

Considering close interactions between sleep, immunity and intestinal inflammation, sleep disorders could be a predictor of flares.

The purpose of this study is to demonstrate that sleep efficacy decreases before IBD flare.

Patients in remission will be assessed for IBD symptoms (activity scores, biological factors) and sleep disorders (actigraphy, DREEM®, questionnaires) during one year.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 and under 65 years of age.
* Patient with Inflammatory Bowel Disease diagnosed for at least 3 months.
* Patient in remission, for at least 3 months:

  1. clinical remission: Harvey-Bradshaw score (HBI) < 5 for CD and a Mayo score < 3 for UC
  2. and biological remission: absence of objective inflammation defined by CRP < 5 mg/L and/or fecal calprotectin < 250 µg/g.
* Patient must sign informed consent form to participate to the study.
* Patient affiliated to or benefiting from a social security plan.

Exclusion Criteria:

* Patient with complications (obstructive symptoms, fistulas or intra-abdominal abscesses in the previous three months).
* Patient with extensive bowel resection (> 40 cm of small bowel).
* Patient with an ileostomy or colostomy.
* Patient diagnosed with sleep disorders.
* Patient without legal capacity to consent.
* Pregnant, parturient or nursing women.
* Persons deprived of liberty by judicial or administrative decision.
* Persons under psychiatric care.
* Persons admitted to a health or social institution for purposes other than research.
* Persons of full age who are subject to a legal protection measure (guardianship, curators).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-04-08 (Estimated); Study Completion 2028-06-08 (Estimated)

PRIMARY OUTCOMES:
rate of relapse | 12 months after baseline
  For Crohn's disease:
  Harvey Bradshaw Index ≥ 5 AND a CRP > 5 mg/L and/or calprotectin > 250 µg/g
  For ulcerative colitis:
  Mayo ≥ 3 AND a CRP > 5 mg/L and/or calprotectin > 250 µg/g Sleep efficiency will be measured by actimetry and expressed as a percentage. Sleep efficiency is defined as the ratio of total time spent asleep compared to total time spent in bed. An actinometer will collect one efficiency measurement per night; an average per week will then be calculated from the daily measurements.

SECONDARY OUTCOMES:
Sleep efficiency calculated by actimetry and expressed in percentage. | 12 months after baseline
  Patient will wear actimeters on the wrist for 1 year continuously.
Intra-sleep wakefulness duration (min), sleep latency (min) and sleep duration (min) | 12 months after baseline
  Intra-sleep wakefulness duration (min), sleep latency (min) and sleep duration (min) will be measured with an actinometer, and averaged per week. Patient will wear actinometers on the wrist for 1 year continuously.
total sleep time | 12 months after baseline
  Sleep parameters evaluated by headband are:
  * sleep macrostructure: concerns the polycyclic organization of sleep and the following quantitative parameters: total sleep time (min), sleep onset latency (min), intra-sleep wake duration (min), polysomnographic sleep efficiency (= total sleep time/time in bed), quantity of different sleep stages (min and % of total sleep time)
  * sleep microstructure: concerns the index of micro-arousals (number/hour) and spindle density (number/minute) or delta spectral power in slow wave sleep (delta/total power ratio).
sleep onset latency | 12 months after baseline
  Sleep parameters evaluated by headband are:
  * sleep macrostructure: concerns the polycyclic organization of sleep and the following quantitative parameters: total sleep time (min), sleep onset latency (min), intra-sleep wake duration (min), polysomnographic sleep efficiency (= total sleep time/time in bed), quantity of different sleep stages (min and % of total sleep time)
  * sleep microstructure: concerns the index of micro-arousals (number/hour) and spindle density (number/minute) or delta spectral power in slow wave sleep (delta/total power ratio).
intra-sleep wake duration | 12 months after baseline
  Sleep parameters evaluated by headband are:
  * sleep macrostructure: concerns the polycyclic organization of sleep and the following quantitative parameters: total sleep time (min), sleep onset latency (min), intra-sleep wake duration (min), polysomnographic sleep efficiency (= total sleep time/time in bed), quantity of different sleep stages (min and % of total sleep time)
  * sleep microstructure: concerns the index of micro-arousals (number/hour) and spindle density (number/minute) or delta spectral power in slow wave sleep (delta/total power ratio).
polysomnographic sleep efficiency | 12 months after baseline
  Sleep parameters evaluated by headband are:
  * sleep macrostructure: concerns the polycyclic organization of sleep and the following quantitative parameters: total sleep time (min), sleep onset latency (min), intra-sleep wake duration (min), polysomnographic sleep efficiency (= total sleep time/time in bed), quantity of different sleep stages (min and % of total sleep time)
  * sleep microstructure: concerns the index of micro-arousals (number/hour) and spindle density (number/minute) or delta spectral power in slow wave sleep (delta/total power ratio).
quantity of different sleep stages | 12 months after baseline
  Sleep parameters evaluated by headband are:
  * sleep macrostructure: concerns the polycyclic organization of sleep and the following quantitative parameters: total sleep time (min), sleep onset latency (min), intra-sleep wake duration (min), polysomnographic sleep efficiency (= total sleep time/time in bed), quantity of different sleep stages (min and % of total sleep time)
  * sleep microstructure: concerns the index of micro-arousals (number/hour) and spindle density (number/minute) or delta spectral power in slow wave sleep (delta/total power ratio).
index of micro-arousals | 12 months after baseline
  Sleep parameters evaluated by headband are:
  * sleep macrostructure: concerns the polycyclic organization of sleep and the following quantitative parameters: total sleep time (min), sleep onset latency (min), intra-sleep wake duration (min), polysomnographic sleep efficiency (= total sleep time/time in bed), quantity of different sleep stages (min and % of total sleep time)
  * sleep microstructure: concerns the index of micro-arousals (number/hour) and spindle density (number/minute) or delta spectral power in slow wave sleep (delta/total power ratio).
spindle density | 12 months after baseline
  Sleep parameters evaluated by headband are:
  * sleep macrostructure: concerns the polycyclic organization of sleep and the following quantitative parameters: total sleep time (min), sleep onset latency (min), intra-sleep wake duration (min), polysomnographic sleep efficiency (= total sleep time/time in bed), quantity of different sleep stages (min and % of total sleep time)
  * sleep microstructure: concerns the index of micro-arousals (number/hour) and spindle density (number/minute) or delta spectral power in slow wave sleep (delta/total power ratio).
delta spectral power in slow wave sleep | 12 months after baseline
  Sleep parameters evaluated by headband are:
  * sleep macrostructure: concerns the polycyclic organization of sleep and the following quantitative parameters: total sleep time (min), sleep onset latency (min), intra-sleep wake duration (min), polysomnographic sleep efficiency (= total sleep time/time in bed), quantity of different sleep stages (min and % of total sleep time)
  * sleep microstructure: concerns the index of micro-arousals (number/hour) and spindle density (number/minute) or delta spectral power in slow wave sleep (delta/total power ratio).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Clermont-Ferrand, Hôpital d'Estaing, Clermont-Ferrand
  - CHU Grenoble Hôpital Michallon-Site Nord, Grenoble
  - Lyon Sud hospital, Pierre-Bénite
  - CHU Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No